CLINICAL TRIAL: NCT06550388
Title: Effect of Brief Lifestyle Interventions on the Subjective Sleep Quality of Patients With Chronic Insomnia
Brief Title: Subjective Sleep Quality of Patients With Chronic Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexa Kane, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-004753
Record Dates: First submitted 2024-07-22; First posted 2024-08-13 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Education (Other): In addition to the traditional course of CBT-I, the PI will recommend patient to increase physical activity minutes per week. The increase in physical activity will be based on patient's current level of physical activity.
  Interventions: Behavioral: Physical Activity
- Nutritional Education (Other): In addition to the traditional course of CBT-I, the PI will provide education and materials regarding the Mediterranean Diet. Patient will be provided with the Mayo Clinic booklet on Mediterranean Diet and asked to increase their daily intake in two categories assessed by the Mini-EAT.
  Interventions: Behavioral: Nutritional Education

INTERVENTIONS:
Behavioral: Nutritional Education — In addition to the traditional course of CBT-I, the PI will provide education and materials regarding the Mediterranean Diet. Patient will be provided with the Mayo Clinic booklet on Mediterranean Diet and asked to increase their daily intake in two categories assessed by the Mini-EAT.
  Arms: Nutritional Education
Behavioral: Physical Activity — In addition to the traditional course of CBT-I, the PI will recommend patient to increase physical activity minutes per week. The increase in physical activity will be based on patient's current level of physical activity.
  Arms: Physical Activity Education

SUMMARY:
The purpose of this study is to assess subjective sleep quality, diet quality, physical activity in patients with chronic insomnia before and after a brief lifestyle intervention during a traditional course of Cognitive Behavioral Therapy for Insomnia (CBT-I)

DETAILED DESCRIPTION:
Chronic insomnia disorder is highly prevalent, occurring in 4% to 22% of the population in the U.S. The consequences of chronic insomnia are significant including mood disorders, work-related and motor vehicle accidents, and overall poor quality of life. Lack of sleep satisfaction, a hallmark of chronic insomnia, is associated with metabolic syndrome, diabetes, hypertension, coronary heart disease and depression1.

Chronic insomnia is predominantly managed with hypnotics and other medications despite the effectiveness of and patient preference for CBT-I. The American College of Physicians (ACP) and the American Academy of Sleep Medicine (AASM) guidelines for management of chronic insomnia recommend all patients receive Cognitive Behavioral Therapy for Insomnia (CBT-I) as first line treatment for chronic insomnia2,3. CBT-I is a structured, nonpharmacological treatment that uses educational, cognitive, and behavioral strategies. Meta-analyses have shown CBT-I is consistently associated with improved sleep quality in chronic insomnia with or without comorbidities4,5. While the strategies associated with CBT-I have been found to be effective for the management of chronic insomnia, lifestyle intervention to improve patients' diet and physical activity is not part of traditional CBT-I. The field of behavioral sleep medicine can expand interventional strategies to promote health and well-being while also optimizing sleep health.

A pathway to improve sleep health is a shift from a typical medicine perspective which emphasizes identification and treatment of symptoms, to a health promotion perspective, which emphasizes the promotion of overall well-being. Incorporating principles from lifestyle medicine and behavioral sleep medicine can both identify and treat sleep disorders plus promote overall health including education regarding diet quality and exercise. Targeting diet quality and physical activity education within the context of CBT-I will underscore the importance of nonpharmacological treatment and the promotion of health and well-being which is central to behavioral sleep and lifestyle medicine.

The etiology of chronic insomnia disorder is multifactorial with research supporting poor diet and lack of physical activity as contributing factors to poor sleep. Previous studies have reported higher diet quality promotes better sleep quality and mental health. Sleep deprivation and sleep disturbances have been linked to poor diet quality. Eating too quickly or skipping meals, overabundant meals, irregular mealtimes, and poor food quality, all are dietary causes of sleep disorders. Additionally, the timing of meals, including frequency and regularity of snacks, may desynchronize circadian rhythm, affect metabolism, and favor obesity6. There is mounting evidence suggesting sleep influences dietary choices as well. Individuals who sleep less are more likely to prefer energy-rich foods (e.g., fats and refined carbohydrates), eat fewer vegetables, and choose irregular eating patterns7.

Additionally, several pathways have been proposed regarding benefits of the Mediterranean diet and healthy dietary patterns on sleep, including the role of the gut microbiome8, inflammation and the consumption of dietary tryptophan and melatonin9. Some observational studies have shown a high intake of fruit and vegetables is associated with better sleep quality and lower risk of insomnia while a cohort study of older adults in Spain showed that higher consumption of red meat was associated with poor sleep quality and snoring10,11.

Recent studies have also highlighted the importance of physical activity and the impact on sleep quality. Low levels of physical activity have been reported as significant risk factors for both prevalent and incident insomnia12. One study documented improvements in sleep after days with more acute moderate-intensity activity in patients diagnosed with chronic insomnia13. Physical activity and sleep likely influence each other in both physiological and psychological pathways. For example, in older adults, increasing physical activity has been shown to improve excessive daytime sleepiness and reduce prevalence of insomnia symptoms14. Although there have been studies assessing the association between sleep quality and physical activity, very little has looked at patients diagnosed with chronic insomnia and we believe this is the first study to add a brief lifestyle intervention to traditional CBT-I.

There is support for the inclusion of healthy diet education and increased physical activity in interventions programs, such as CBT-I, to improve sleep quality among individuals diagnosed with chronic insomnia. Combining health promoting behaviors in conjunction with CBT-I is likely to be of great importance in preventing a large set of chronic non-communicable disease. At the very least, the combination of traditional CBT-I with healthy diet education and physical education may increase sleep quality, diet quality and physical activity for patients diagnosed with chronic insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Insomnia
* 18-70 years of age

Exclusion Criteria:

* Known untreated sleep disorder
* Cardiovascular diagnosis that would not allow safe increase of physical activity
* Diabetes
* Pregnancy or lactation
* Current use of a vegan diet or Mediterranean diet
* BMI ≤ 22
* Score higher than 15 on PHQ-8
* Diagnosed with a severe neurological or sensory impairment that would significant impact participation
* Currently performing shift work/diagnosis of a circadian rhythm disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in sleep quality measured by the Pittsburgh Sleep Quality Index | Baseline, 84 days
  Measures the severity of sleep disturbances. Possible scores range from 0 to 21 with higher scores indicating a worse outcome/more severe symptoms of sleep disturbance.

SECONDARY OUTCOMES:
Change in insomnia measured by the Insomnia Severity Index | Baseline, 14 days, 28 days, 42 days, 56 days, 70 days, 84 days
  Self-reported insomnia severity index questionnaire score, using a total score, scale of 0-7 is no clinically significant insomnia, 8-14 is subthreshold insomnia, 15-21 is clinical insomnia (moderate severity), 22-28 is Clinical insomnia (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Kane, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No